CLINICAL TRIAL: NCT04911049
Title: Prevalence and Pathophysiology of Systemic Arterial Pressure Abnormalities in Childhood Sickle Cell Disease
Acronym: DrépaPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201318
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; systemic hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood Pressure measurement — Blood Pressure measurement

SUMMARY:
It is usually found that the blood pressure of adults with sickle cell disease is lower than in non-sickle cell patients. On the other hand, three recent prospective studies in children with sickle cell disease show prevalence of hypertension diagnosed by ambulatory blood pressure measurement (ABPM) ranging from 32 to 45% but on small numbers of patients (n = 54 at most). This hypertension appears to affect kidney function and has been previously associated with the risk of hemorrhagic stroke. It is therefore important to know the prevalence of hypertension in children with sickle cell disease and to determine its mechanisms. The factors which could explain this high prevalence are the increase in arterial stiffness and the increase in systemic vascular resistance linked to the alteration of the sympathovagal balance contributing to the regulation of vascular tone. Indeed, a disturbance of this balance with an increase in vasoconstrictor sympathetic tone has already been found. Hypothesis: In a subgroup of sickle cell children there is systemic hypertension (prevalence: main objective) linked to the alteration of the sympathovagal balance already established during sickle cell disease (increase in sympathetic tone and decrease in parasympathetic tone) affecting systemic vascular resistance (secondary pathophysiological objectives).

DETAILED DESCRIPTION:
Main objective (200 children): To evaluate the prevalence of elevated blood pressure (former pre-hypertension) and hypertension (including masked hypertension) in children with sickle cell disease. Secondary objectives (60 children): to evaluate the prevalence of loss of nocturnal decrease in blood pressure (dipping); to evaluate arterial stiffness (pulse wave velocity: PWV) and vascular resistance (Augmentation Index, AI) in the different groups: normal, pre-hypertension and hypertension; to evaluate the cardiac sympathovagal balance by studying heart rate variability (HRV) in the three groups: normal, pre-hypertension and hypertension; to evaluate arterial in the three groups: normal, pre-hypertension and hypertension; to evaluate whether the absence of nocturnal dipping is or is not an associated factor of abnormal arterial stiffness, systemic vascular resistance, sympathovagal balance or baroreflex by comparison of subjects with normal dipping versus abnormal dipping.

ELIGIBILITY:
Inclusion Criteria:

* child (age <18 years);
* sub-Saharan or Caribbean origin;
* major sickle cell disease (SS, SC and Sbeta-thalassemia);
* height ≥ 120 cm; absence of treated hypertension or antihypertensive treatment;
* parents informed and not opposed to participation in research

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: childhood sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring (ABPM) | 2 years
  mean, systolic and diastolic arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère KOEHL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bokov P, Koehl B, Benzouid C, Verlhac S, Missud F, Benkerrou M, Delclaux C. No Increase in Masked Hypertension Prevalence in Children With Sickle Cell Disease in France. Am J Hypertens. 2024 Apr 15;37(5):358-365. doi: 10.1093/ajh/hpae013. PMID 38323455